CLINICAL TRIAL: NCT02350127
Title: Preventing Loss of Independence Through Exercise (PLIE) in Persons With Dementia
Acronym: PLIE-VA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: LifeLong Marin Adult Day Health Center (Other); Institute on Aging, San Francisco, CA (Other); Catholic Charities (Other); Alzheimer's Services of the East Bay (Other); Bayview Hunters Point Adult Day Health Center (Other); Primrose Alzheimer's Living, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: D1507-I; 5I01RX001507-02 (NIH)
Record Dates: First submitted 2015-01-16; First posted 2015-01-29 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: dementia; clinical trial; behavioral intervention; exercise; complementary and alternative medicine; cognition; function; quality of life
MeSH Terms: conditions — Dementia; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Start (Experimental): The Immediate Start group will participate in the Preventing Loss of Independence through Exercise (PLIE) group movement program for 1 hour, 2-3 days/week, for 4 months. After the intervention has been completed, they will be encouraged to maintain PLIE activities on their own for the next 4 months.
  Interventions: Behavioral: Preventing Loss of Independence through Exercise (PLIE); Behavioral: Usual Care
- Delayed Start (Active Comparator): Study participants who are randomized to the Delayed Start control group will be placed on a waitlist and will be encouraged to continue participating in their usual activities at the adult day center or in their community setting for 4 months. After the 4-month waitlist period ends, they will participate in the PLIE program for 1 hour, 2-3 days/week, for 4 months.
  Interventions: Behavioral: Preventing Loss of Independence through Exercise (PLIE); Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Preventing Loss of Independence through Exercise (PLIE) — PLIE is an integrative group movement program that focuses on training procedural memory for the ability to perform the movements that are most needed for daily function (e.g., transitioning safely between sitting and standing) while increasing mindful body awareness and encouraging social connection. It combines elements from a wide range of Eastern and Western exercise modalities, including occupational therapy, physical therapy, yoga, tai chi, Feldenkrais, Rosen Method, dance movement therapy and mindfulness meditation.
Behavioral: Usual Care — Usual care activities will vary between participants. Some will be attending the adult day center and may be engaging in structured physical, mental and/or social activities. Other participants will be living in the community and may engage in physical, mental, and/or social activities on their own or with a caregiver.

SUMMARY:
Nearly 1 in 10 older Veterans have dementia, which is a devastating condition that leads to a progressive loss of independence and functional status. Currently available dementia medications do not alter the disease course. Therefore, it is critically important to identify effective strategies for helping older Veterans living with dementia to enhance their functional status and quality of life. The investigators have developed a novel, integrative group movement program called Preventing Loss of Independence through Exercise (PLIE) that incorporates elements from Eastern and Western exercise modalities and is designed to build and maintain the capacity to perform basic functional movements while increasing mindful body awareness and enhancing social connection. Pilot study results suggested that PLIE is associated with meaningful improvements in physical function, cognitive function and quality of life as well as reduced caregiver burden. The goal of the current study is to perform a full-scale randomized, controlled trial to test the efficacy of PLIE in older Veterans with dementia.

DETAILED DESCRIPTION:
The goal of the proposed study is to perform a randomized, controlled trial (RCT) to test the efficacy of a novel integrative group movement program called Preventing Loss of Independence through Exercise (PLIE) on function and quality of life in older Veterans living in the community with dementia. Dementia is a devastating condition that affects nearly 1 in 10 older Veterans (~1 million individuals). Current dementia medications have minimal impact on function and quality of life and do not stop or slow the disease course; however, there is growing evidence that behavioral interventions such as exercise have a variety of beneficial effects in individuals with dementia. PLIE was developed based on recent discoveries in neuroscience and experimental psychology that have found that, although explicit memory (the ability to consciously recall new information) is impaired in individuals with dementia, implicit memory (unconscious learning that typically occurs through repeated exposure) is relatively preserved. Therefore, PLIE focuses on training procedural memory (unconscious learning of procedures) to build the strength and capacity to perform the movements that are most needed for daily function (e.g., transitioning safely from sitting to standing). In addition, to maximize the benefits of the training, PLIE integrates elements of Eastern and Western exercise modalities to develop mindful body awareness and enhance social connection. The investigators completed a pilot study of the PLIE program at an adult day center in San Francisco, CA, finding that it was associated with clinically meaningful improvements in cognitive function, physical performance and quality of life as well as reduced caregiver burden when compared with usual care at the facility. The current study will enable the investigators to build on these pilot study results by performing a full-scale RCT at adult day centers in Northern California. Most VA Medical Centers currently contract with community-based organizations to provide adult day care to eligible Veterans with dementia. Therefore, sites for the current study will be adult day centers that have current contracts with local VA medical centers. Within each center, study participants will be randomly assigned to receive the PLIE intervention program (1 hour, 2-3 days/week, 4 months) or Usual Care (UC) control (standard center activities, 1 hour, 2-3 days/week, 4 months) (N=120, 60/group) using a waitlist design. The co-primary outcomes are 4-month change in physical function (Short Physical Performance Battery, SPPB), cognitive function (Alzheimer's Disease Assessment Scale - cognitive subscale, ADAS-cog) and quality of life (Quality of Life in Alzheimer's Disease, QOL-AD). Changes in caregiver feelings (Caregiver Burden Inventory, CBI; Positive Aspects of Caregiving, PAC), mood (Geriatric Depression Scale, GDS), fear of falling (Falls Efficacy Scale, FES), independence (Disability Assessment for Dementia, DAD) and dementia-related behaviors (Neuropsychiatric Inventory, NPI) will be examined as secondary outcomes. To account for the waitlist design, all outcomes will be assessed at baseline, 4 months and 8 months. The proposed project will address a critically important Veterans' health problem related to optimizing functional status and quality of life in older Veterans with dementia. It is directly responsive to Request for Applications (RFA) RX-14-011 (RR&D Merit Review Award for Research on Amyotrophic Lateral Sclerosis, Parkinson's Disease and Alzheimer's Disease), which has identified "pioneering new and innovative rehabilitation methodologies to restore function and improve quality of life for Veterans living with [these] neurodegenerative diseases" as a "major focus." Many patients and caregivers currently feel that little is being done to help individuals with dementia maintain function and quality of life. The current study will utilize rigorous research methods to test the efficacy of an innovative and promising new program for older adults with dementia. If the program is successful, the investigators will work with VA and community-based organizations to implement PLIE more broadly.

ELIGIBILITY:
Inclusion Criteria:

* 120 dyads of individuals with dementia and their primary caregivers will be enrolled, with a goal of 20 dyads per intervention site.
* Veterans with dementia will be prioritized for enrollment at each site.
* Enrollment will be opened to non-Veterans with dementia at the site if there are not an adequate number of Veterans to fill the group.
* Caregivers are not required to be Veterans, but their participation is necessary because they are providing care to the primary participants, many of whom will be Veterans.

Inclusion criteria, primary participant:

* diagnosis of memory loss or dementia
* mild to moderate severity (defined as Clinical Dementia Rating of 0.5, 1 or 2)
* English language fluency
* attendance or willingness to attend adult day health center at least 2 days/week on days that PLIE will be offered

Inclusion criteria, caregivers:

* Provide care for primary participant
* Able to answer study questionnaires related to participant's functional status, dementia-related behaviors, quality of life and their own burden.
* English language fluency

Exclusion Criteria:

Exclusion criteria, primary participant:

* Plans to change days of attendance during the study period so that participant would no longer be attending on at least 2 PLIE days/week.
* Planning to leave the facility during the study period and not willing to come for PLIE classes at least 2 days/week
* Severe vision or hearing impairment (e.g., unable to see or hear well enough to follow instructions)
* Several physical impairment (e.g., paralysis or hemi-paralysis; wheel-chair or bed bound)
* Severe mental health condition (e.g., uncontrolled depression, PTSD, bipolar disorder)
* Limited life expectancy (e.g., enrolled in or eligible for hospice; metastatic cancer)
* Started dementia medication (cholinesterase inhibitor or memantine) in past 3 months.
* Planning to change dementia medication during the study period
* Current participation in another research study
* Lack of legally authorized representative to provide consent
* Lack of consent/assent to study procedures

Exclusion criteria, caregivers:

* Severe vision or hearing impairment (e.g., unable to see or hear well enough to follow instructions)
* Several physical impairment (e.g., paralysis or hemi-paralysis; wheel-chair or bed bound)
* Severe mental health condition (e.g,. uncontrolled depression, PTSD, bipolar)
* Limited life expectancy (e.g., enrolled in or eligible for hospice; metastatic cancer)
* lack of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-05-04 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Barnes, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes DE, Mehling W, Wu E, Beristianos M, Yaffe K, Skultety K, Chesney MA. Preventing loss of independence through exercise (PLIE): a pilot clinical trial in older adults with dementia. PLoS One. 2015 Feb 11;10(2):e0113367. doi: 10.1371/journal.pone.0113367. eCollection 2015. PMID 25671576
- [Background] Wu E, Barnes DE, Ackerman SL, Lee J, Chesney M, Mehling WE. Preventing Loss of Independence through Exercise (PLIE): qualitative analysis of a clinical trial in older adults with dementia. Aging Ment Health. 2015;19(4):353-62. doi: 10.1080/13607863.2014.935290. Epub 2014 Jul 14. PMID 25022459
- See also: Facebook page for PLIE program — https://www.facebook.com/plie4dementia
- See also: Osher Center description of PLIE program — http://www.osher.ucsf.edu/research/current-research/preventing-loss-of-independence-through-exercise-plie/
- See also: SFVA link to ongoing research studies — http://www.sanfrancisco.va.gov/research/study.asp

RESULTS

PARTICIPANT FLOW:
Period: 4-Month Assessment
Arm/Group | Immediate Start | Delayed Start
Started | 44 | 44
Completed Baseline | 42 (Withdrew prior to baseline due to time constraints (n=1) and lack of interest (n=1)) | 43 (Withdrew prior to baseline due to health issue (n=1))
Completed | 33 | 35
Not Completed | 11 | 9
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Death | 1 | 0
Period: 8-Month Assessment
Arm/Group | Immediate Start | Delayed Start
Started | 33 | 35
Completed | 27 | 26
Not Completed | 6 | 9
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Start | Delayed Start | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.0 (7.8) | 79.0 (7.3) | 79.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 30 | 29 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 38 | 38 | 76
  Race/Ethnicity: Asian | 3 | 1 | 4
  Race/Ethnicity: Black/African American | 3 | 1 | 4
  Race/Ethnicity: Native Hawaiian/Pacific Islander | 0 | 1 | 1
  Race/Ethnicity: Hispanic/Latino (any race) | 0 | 2 | 2
  Race/Ethnicity: Multiple/Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 44 | 44 | 88
Participant MOCA Score [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment (MOCA) is a standard measure of global cognitive function in which scores may range from 0 to 30 with higher scores indicating better cognitive function and scores less than 26 indicating cognitive impairment. Population: The MOCA was administered immediately after obtaining informed consent and was missing for 2 participants. The baseline assessment was typically performed at a separate visit. Some participants withdrew after consenting but before completing the baseline assessment, and their scores are included.
  units on a scale
    number analyzed (Participants) | 43 | 43 | 86
    (all) | 10.7 (7.3) | 13.8 (6.9) | 12.3 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Scale in Alzheimer's Disease (QOL-AD)
Description: The Quality of Life Scale in Alzheimer's Disease (QOL-AD) is a standard quality of life measure that asks parallel questions of affected individuals and caregivers. Current quality of life is rated as poor (1 point), fair (2 points), good (3 points) or excellent (4 points) in 13 areas: physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores around the house, ability to do things for fun, money, and life as a whole. Scores may range from 13 to 52 with higher scores reflecting better quality of life. Prior studies have found that the QOL-AD is a valid and reliable measure, with Cronbach's alpha of 0.84 for patient reports and 0.86 for caregiver reports and interrater reliability based on Cohen's kappa values >0.70.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 42 | 43
score on a scale | 38.8 (6.2) | 40.0 (4.3)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; adjusted for participant baseline MOCA, robust VCE; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Final Values) = 1.79, 95% CI 2-sided [-0.59 to 4.18], Standard Error of Mean 1.22
Statistical Analysis 2: Comparison: Immediate Start vs Delayed Start; restricted to completers; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [0.2 to 5.6], Standard Error of Mean 1.4

2. Primary Outcome: Short Physical Performance Battery (SPPB)-Modified
Description: The SPPB was developed by the National Institute on Aging to provide an objective tool for measuring physical performance in older adults. Lower body strength is assessed based on time to complete 5 chair stands without using arms. Balance is assessed based on the ability to hold different stands for 10 seconds, including the side-by-side, semi-tandem and full tandem stands. Mobility is assessed based on usual walking speed over a 3-meter walking course. The total SPPB score is the sum of the 3 component scores and may range from 0 to 12. Higher scores reflect better performance.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 42 | 43
score on a scale | 6.1 (3.0) | 6.1 (3.2)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.68, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-1.23 to 0.80], Standard Error of Mean 0.52 — Adjusting for baseline participant MOCA scores, robust vce

3. Primary Outcome: Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog)
Description: The Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog) is one of the most commonly used outcome measures in dementia drug treatment trials and is one of the measures considered by the Food and Drug Administration for approval of dementia medications. It includes direct assessment of learning (10-word list), naming (objects), following commands, constructional praxis (figure copying), ideational praxis (mailing a letter), orientation (person, time, place), recognition memory and remembering test instructions. Scores may range from 0 to 70 with higher scores reflecting worse cognitive function. Prior studies have found the ADAS-cog to be valid and reliable with Cronbach's alpha greater than 0.8 and test-retest reliability above 0.9.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 42 | 43
score on a scale | 36.7 (13.8) | 30.4 (13.2)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; adjusting for baseline participant MOCA, robust VCE; Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-3.09 to 2.08], Standard Error of Mean 1.32

4. Secondary Outcome: Caregiver Burden Inventory (CBI)
Description: The Caregiver Burden Inventory (CBI) is a standard measure that includes 24 items and 5 domains. Caregivers are asked to rate how often each statement describes their feelings (never, rarely, sometimes, quite frequently, nearly always). The total score may range from 0 to 96 with higher scores reflecting greater feelings of burden.
Time Frame: 4 months
Population: Data missing for 1 immediate start participant (did not have a caregiver) and 1 delayed start participant (did not have a caregiver).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 41 | 42
score on a scale | 31.8 (14.9) | 32.0 (14.9)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.02, Mixed Models Analysis; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [0.8 to 9.4], Standard Error of Mean 2.2

5. Secondary Outcome: Disability Assessment for Dementia (DAD)
Description: The Disability Assessment for Dementia (DAD) is a standard measure of functional independence that asks caregivers whether the participant performed 17 basic and 23 instrumental activities of daily living over the past 2 weeks without reminder or assistance. Each item is rated as yes, no, or not applicable (i.e., never performed, no opportunity to perform). The score reflects the percent of items performed independently, excluding those that were not applicable. Therefore, scores may range from 0 to 100 with higher scores reflecting greater independence. The DAD has high established validity and high test-retest reliability (ICC, 0.96), inter-rater reliability (ICC, 0.95) and internal consistency (Cronbach's alpha, 0.96).
Time Frame: 4 months
Population: Baseline data missing for 2 immediate start participants (1 did not have a caregiver, 1 caregiver did not complete questionnaire) and 1 delayed start participant (did not have a caregiver).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 40 | 42
score on a scale | 52.3 (24.1) | 65.5 (23.9)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.47, Mixed Models Analysis; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-5.4 to 11.6], Standard Error of Mean 4.3

6. Secondary Outcome: Neuropsychiatric Inventory - Number (NPI-N)
Description: The NPI assesses the frequency, severity and level of distress caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and appetite/eating). The NPI-N counts the number of symptoms present. Scores may range from 0 to 12 with higher scores reflecting worse outcomes (i.e., more symptoms).
Time Frame: 4 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 41 | 42
score on a scale | 4.0 (2.8) | 3.5 (2.6)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.1 to 1.1], Standard Error of Mean 0.54

7. Secondary Outcome: Neuropsychiatric Inventory - Frequency*Severity (NPI-FS)
Description: The Neuropsychiatric Inventory - Frequency*Severity subscale (NPI-FS) assesses the frequency and severity of 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and appetite/eating) by caregiver report. NPI-FS was calculated by multiplying the frequency*severity of behaviors, which had a range of 0-144. Higher scores indicate worse outcomes (greater frequency/severity).
Time Frame: 4 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 41 | 42
score on a scale | 15.9 (18.4) | 14.1 (15.9)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.98, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-7.4 to 7.2], Standard Error of Mean 3.7

8. Secondary Outcome: Neuropsychiatric Inventory - Caregiver Distress
Description: Measure of caregiver distress associated with 12 common dementia-related behaviors. Scores may range from 0 to 60 with higher scores reflecting greater distress.
Time Frame: 4 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 41 | 42
score on a scale | 8.1 (8.4) | 8.3 (7.6)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.80, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-2.5 to 3.3], Standard Error of Mean 1.5

9. Secondary Outcome: Quality of Life in Alzheimer's Disease - CG Report About Participant
Description: Caregiver assessment of participant's quality of life. Scores may range from 13 to 52, with higher scores reflecting better quality of life.
Time Frame: 4 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 41 | 42
score on a scale | 31.2 (5.6) | 33.1 (5.1)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.38, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-3.1 to 1.2], Standard Error of Mean 1.1

10. Secondary Outcome: Geriatric Depression Scale (GDS)
Description: Depressive symptoms were assessed in caregivers based on self-report using the GDS - short form, a 15-item yes/no scale. Scores may range from 0 to 15, with higher scores reflecting greater depressive symptomatology.
Time Frame: 4 months
Population: Data missing for 2 immediate start participants (1 did not have a caregiver, 1 did not complete questionnaire) and 1 delayed start participant (did not have a caregiver).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 40 | 42
score on a scale | 3.3 (3.2) | 3.3 (3.0)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.075, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.7 to 0.1], Standard Error of Mean 0.45

11. Secondary Outcome: Positive Aspects of Caregiving (PAC)
Description: A standard measure that asks caregivers to rate their agreement/disagreement with 11 statements about positive aspects of caregiving on a 5-point likert scale (disagree a lot ... agree a lot). Total scores range from 11 to 55 with higher scores indicating more positive feelings
Time Frame: 4 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 41 | 42
score on a scale | 36.9 (8.2) | 39.5 (9.5)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.35, Mixed Models Analysis; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-1.7 to 5.0], Standard Error of Mean 1.7

12. Secondary Outcome: Chair Stand Time
Description: Time to complete 5 chair stands without using arms in seconds. Higher scores reflect worse (slower) performance.
Time Frame: 4 months
Population: Data missing for 10 immediate start and 13 delayed start participants (unable to complete test)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 32 | 30
seconds | 17.7 (8.4) | 18.2 (9.8)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.35, Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-6.1 to 2.1], Standard Error of Mean 2.1

13. Secondary Outcome: Balance Score
Description: From Short Physical Performance Battery, including side-by-side, semi-tandem, and tandem balance. Score may range from 0 to 4, with higher scores indicating better balance.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 42 | 43
score on a scale | 2.4 (1.4) | 2.4 (1.4)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.54, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.8], Standard Error of Mean 0.3

14. Secondary Outcome: Usual Gait Speed
Description: From Short Physical Performance Battery, better of two times in seconds. Higher scores reflect worse (slower) performance.
Time Frame: 4 months
Population: Data missing for 1 delayed start participant (unable to complete test).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 42 | 42
seconds | 5.6 (3.9) | 5.6 (4.2)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.69, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.5 to 2.2], Standard Error of Mean 0.9

15. Secondary Outcome: Timed Up & Go
Description: Measure of mobility in which participant is timed while standing up from a seated position, walking around a cone that is 8 feet away, and returning to a seated position. Higher scores reflect worse (slower) performance.
Time Frame: 4 months
Population: Data missing for 2 immediate start and 3 delayed start participants (unable to complete test).
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 40 | 40
seconds | 15.7 (10.8) | 16.1 (18.1)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.88, Mixed Models Analysis; Median Difference (Final Values) = -0.8, 95% CI 2-sided [-10.9 to 9.3], Standard Error of Mean 5.2

16. Secondary Outcome: Sit & Reach
Description: Measure of flexibility in which participant reaches toward toes with a straight leg. Score reflect closest to touching, with positive values reflecting past toes and negative values reflecting not touching toes.
Time Frame: 4 months
Population: Data missing for 3 immediate start and 2 delayed start participants (unable to complete test).
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 39 | 41
inches | -4.3 (5.0) | -4.0 (4.2)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.26, Mixed Models Analysis; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.7 to 2.5], Standard Error of Mean 0.8

17. Secondary Outcome: Falls Efficacy Scale (FES) - Participant Report
Description: A standard measure of falls efficacy that can be administered to people with cognitive impairment or caregivers and asks about concern about the possibility of falling doing 10 daily tasks (e.g., taking a bath or shower) on a 4-point likert scale (not at all, somewhat, fairly or very concerned). Scores may range from 10 to 40 with higher scores reflecting worse outcomes (i.e., greater concern about falling).
Time Frame: 4 months
Population: Data missing for 1 immediate start and 1 delayed start participants (unable to answer questions).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Start | Delayed Start
Number analyzed (Participants) | 41 | 42
score on a scale | 14.2 (6.7) | 14.1 (5.3)
Statistical Analysis 1: Comparison: Immediate Start vs Delayed Start; Test type: Superiority; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.9 to 0.2], Standard Error of Mean 1.1

18. Post Hoc Outcome: Satisfaction Score
Description: Caregivers were sent an anonymous satisfaction survey after completion or withdrawal with a pre-paid return envelope. Satisfaction was rated on a 5-point Likert scale (1=Highly Unsatisfied to 5=Highly Satisfied). Open-ended questions asked about changes observed in study participants and themselves when participating in the program, what they liked the most and found most challenging, and other comments. Qualitative content analyses were performed to identify key domains and sub-domains described.
Time Frame: 8 months
Population: 47 of 88 (53%) caregivers returned the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Evaluation Group Respondents: All caregivers were sent an anonymous evaluation survey with a pre-paid return envelope upon study completion or withdrawal.
Arm/Group | Evaluation Group Respondents
Number analyzed (Participants) | 47
score on a scale | 4.5 (0.9)

ADVERSE EVENTS:
Time Frame: 8 months
Description: Adverse events were collected systematically in both groups during monthly check-in calls by asking caregivers whether study participants had experienced any major health-related events since the last contact. In addition, research staff logged adverse events that they learned about during other interactions with study participants. Adverse events were classified as serious (death, hospitalization, persistent disability, life-threatening) or not serious and were not classified by organ system.
Arm/Group | Immediate Start | Delayed Start
All-Cause Mortality (participants affected / at risk) | 2/44 | 1/44
Serious Adverse Events (participants affected / at risk) | 8/44 | 10/44
Other Adverse Events (participants affected / at risk) | 20/44 | 12/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start (N=44) | Delayed Start (N=44)
Hospitalization (General disorders) | 6 (7) | 8 (10) — Any hospitalization
Life-threatening (General disorders) | 2 (2) | 2 (2) — Decline in health status, stroke, myocardial infarction
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start (N=44) | Delayed Start (N=44)
Not serious (General disorders) | 15 (30) | 10 (21)
Other AE (General disorders) | 7 (8) | 2 (3) — ER/urgent care visit, fall/fracture, major life event
Procedures (General disorders) | 1 (1) | 0 (0) — Surgery

LIMITATIONS AND CAVEATS:
Final enrollment lower than planned due to: 1) unexpected study site relocation and 2) enrollment difficulty at one study site. In addition, withdrawal was higher than anticipated primarily due to declining health status unrelated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT02350127/Prot_SAP_000.pdf